CLINICAL TRIAL: NCT07177196
Title: An Open-label Single Center Study of an Individualized Antisense Oligonucleotide Treatment for Retinal Dystrophy Associated With a Pathogenic PRPH2 Variant
Brief Title: Personalized Antisense Oligonucleotide Therapy for a Single Participant With PRPH2 Mutation Associated With Retinal Dystrophy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: n-Lorem Foundation (Other)
Collaborators: University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 812793
Record Dates: First submitted 2025-09-02; First posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Retinal Dystrophy
MeSH Terms: conditions — Retinal Dystrophies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental)
  Interventions: Drug: nL-PRPH2-001

INTERVENTIONS:
Drug: nL-PRPH2-001 — Personalized antisense oligonucleotide

SUMMARY:
This research project entails delivery of a personalized antisense oligonucleotide (ASO) drug designed for a single participant with Retinal Dystrophy due to PRPH2 mutation

DETAILED DESCRIPTION:
This is an interventional study to evaluate the safety and efficacy of treatment with an individualized antisense oligonucleotide (ASO) treatment in a single participant with Retinal Dystrophy due to PRPH2 mutation

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of retinal dystrophy as a result of the PRPH2 variant
* Have written informed consent (signed and dated), and able to comply with all study requirements, and any authorization required by local law
* Be able to travel to the study site and adhere to study related follow-up examinations and/or procedures
* Have a molecular diagnosis of a heterozygous PRPH2 variant: c.623G>A (p.Gl208Asp) based on genetic testing at Screening (a historic genetic testing report from a certified laboratory is acceptable with Sponsor/Investigator approval)
* Have a BCVA in the worse eye of at least Count Fingers (CF) or better
* Have clear ocular media and adequate pupillary dilation to permit good quality retinal imaging, as determined by the Investigator
* Be a non-pregnant and non-lactating female, and either surgically sterile (e.g., ≥6 weeks post bilateral salpingectomy, bilateral oophorectomy with or without hysterectomy, tubal ligation) or post-menopausal (12 months of spontaneous amenorrhea in females >55 years of age or, in females < 55 years, have had 12 months of spontaneous amenorrhea without alternative medical cause); male participants and their female partners of childbearing potential must use appropriate contraception methods, or refrain from sexual activity for the duration of the study and for 3 months after the last study treatment; for women of childbearing potential for whom the Investigator considers that the potential benefit outweighs any risk to the unborn fetus, a highly effective method of contraception must be used

Exclusion Criteria:

* There is any condition that in the opinion of the Investigator, would ultimately prevent the participant from completion of the study procedures
* There is a present (current) active ocular infection (including herpes simplex virus, varicella zoster or cytomegalovirus) in either eye
* There is current cystoid macular edema (CME) in the treatment eye(s); CME is permissible if stable for 3 months in the opinion of the Investigator (with or without treatment); past CME is permissible if resolved for more than 1 month
* There are lens opacities in the eye(s) to be treated that are clinically significant in the opinion of the Investigator or that would prevent clinical and photographic evaluation of the retina
* Receipt within 1 month prior to informed consent of any intraocular or periocular surgery, or IVT injection, or planned/anticipated intraocular surgery or procedure during the course of the study
* There is current use of, or treatment within the past 3 months or planned treatment of drugs known to be toxic to the lens, retina or optic nerve including but not limited to systemic/intraocular steroids, amiodarone, desferriosamine/desferoxamine, chloroquine/hydroxychloroquine sulfate (Plaquenil), tamoxifen, ethambutol, phenothiazine derivatives including chlorpromazine, fluphenazine (deconoate) levomepromazine, and thioridazine; intermittent use of intraocular steroids may be considered for inclusion following approval by the Investigator
* Any prior receipt of genetic or stem-cell therapy for ocular or non-ocular disease
* There is any secondary or alternate genetic cause of retinal disease other than the heterozygous PRPH2 c.623G>A (p.Gly208Asp) variant
* There has been use of any investigational drug or device within 3 months or 5 half-lives of the first treatment day (Day 1), whichever is longer, or plans to participate in another study of a drug or device during the trial period and for 3 months after the end of the trial period
* There is presence of any significant ocular/non-ocular disease/disorder (including laboratory abnormalities) which, in the opinion of the Investigator, may put the participant at risk, or may influence the results of the trial, or impact the ability of the participant to participate in the trial
* The intraocular pressure in the eye(s) to be treated is greater than 25 mmHg (even in the presence of glaucoma or ocular hypertension which is stabilized on therapy)
* Prior pars plana vitrectomy in the eye(s) to be treated that may affect treatment in the opinion of the Investigator
* Presence of any intravitreal device (e.g., steroid implant)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2025-08-28 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability | Baseline to 24 months
  Incidence and severity of treatment emergent ocular adverse events (TEAEs) and serious ocular adverse events
Safety and Tolerability | Baseline to 24 months
  Incidence and severity of non-ocular TEAEs and Serious non-ocular adverse events
Safety and Tolerability | Baseline to 24 months
  Change from baseline to Best Corrected Visual Acuity (BCVA) and Low Luminance Visual Acuity (LLVA) as measured at every visit
Safety and Tolerability | Baseline to 24 months
  Change in Slit-lamp biomicroscopy including intraocular pressure (IOP), and dilated indirect ophthalmoscopy
Safety and Tolerability | Baseline to 24 months
  Change in full field electroretinograophy (ffERG) results as measured by electrical activity in the retina
Safety and Tolerability | Baseline to 24 months
  Incidence of treatment emergent abnormalities in safety labs
Safety and Tolerability | Baseline to 24 months
  Incidence of treatment emergent abnormalities in physical exams
Safety and Tolerability | Baseline to 24 months
  Incidence of treatment emergent abnormalities in vital signs

SECONDARY OUTCOMES:
Structure and Function | Baseline to 24 months
  Change from baseline in Spectral domain - Optical Coherence Tomography (SD-OCT)
Structure and Function | Baseline to 24 months
  Change in dilated fundus photography
Structure and Function | Baseline to 24 months
  Change in ultra-widefield fundus autofluorescence (UWF-FAF and Heidelberg FAF)
Structure and Function | Baseline to 24 months
  Change in visual field testing (microperimetry)
Structure and Function | Baseline to 24 months
  Change in participant's visual quality of life as measured by NEI VFQ-25
Structure and Function | Baseline to 24 months
  Change in Best Corrected Visual Acuity (BCVA)

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Undecided